CLINICAL TRIAL: NCT03765788
Title: A Randomized, Parallel-group, Double-blind, Placebo-controlled, Multicenter Phase 2 Trial to Investigate the Safety and Efficacy of Secukinumab (AIN457) in Patients With Giant Cell Arteritis (TitAIN)
Brief Title: A Placebo-controlled Phase 2 Trial to Investigate the Safety and Efficacy of Secukinumab in Giant Cell Arteritis
Acronym: TitAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457ADE11C; 2018-002610-12 (EudraCT Number)
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Giant Cell Arteritis
Keywords: GCA; ain457; Secukinumab; Subcutaneous; Vessel Inflammation; corticosteroid tapering; newly diagnosed or relapsing giant cell arteritis; prednisolone taper regimen; "escape"
MeSH Terms: conditions — Giant Cell Arteritis | interventions — secukinumab; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Participants received secukinumab at a dose of 300 milligrams (mg) as subcutaneous (s.c.) injection at Baseline, Week 1,2,3,4 and then every 4 weeks thereafter through to week 48 along with a 26-week prednisolone tapering regimen.
  Interventions: Drug: Secukinumab 300 mg, s.c.; Drug: Prednisolone
- Placebo (Placebo Comparator): Participants received placebo as subcutaneous (s.c.) injection at Baseline, Week 1,2,3,4 and then every 4 weeks thereafter through to week 48 along with a 26-week prednisolone tapering regimen.
  Interventions: Drug: Prednisolone; Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab 300 mg, s.c. — Secukinumab 300 mg was administered by subcutaneous (s.c.) injections using 1 mL pre-filled syringes (PFSs) throughout the study.
  Other Names: AIN457
  Arms: Secukinumab
Drug: Prednisolone — Prednisolone was provided as tablets (1 mg, 5 mg, 10 mg, 20 mg tablets) for daily administration as tapered regimen from a dose of 25 mg to 60 mg at Baseline to 1 mg at Week 26 (last dose)
Drug: Placebo — Placebo 300 mg was administered by subcutaneous (s.c.) injections using 1 mL pre-filled syringes (PFSs) throughout the study.
  Arms: Placebo

SUMMARY:
This study was designed to evaluate the efficacy and safety of secukinumab compared to placebo to maintain disease remission up to 28 weeks including corticosteroid tapering, as well as up to 1 year (52 weeks) in patients with newly diagnosed or relapsing giant cell arteritis (GCA) who were naïve to biological therapy.

DETAILED DESCRIPTION:
This randomized, parallel-group, double-blind, placebo-controlled, multicenter, Phase II study was designed to evaluate the efficacy of secukinumab compared to placebo in combination with a 26-week prednisolone taper regimen in terms of sustained remission in patients with newly diagnosed or relapsing Giant Cell Arteritis (GCA) who were naïve to biological therapy. The study consisted of a Screening Period of up to 6 weeks (maximum duration), a 52-week Treatment Period and an 8-week Safety Follow-up Period

Patients who did not achieve remission by Week 12, experienced a flare after remission or could not adhere to the prednisolone taper regimen entered "escape". Upon entering "escape", patients received prednisolone at a dose determined by the physician's clinical judgment and continued to receive secukinumab or placebo in a blinded manner.

Safety evaluation was included in all visits including two safety follow-up visits performed 8 and 12 weeks after the last study drug administration.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of GCA classified according to the following criteria:

* Age at onset of disease ≥ 50 years.
* History of ESR ≥ 30 mm/hr or CRP ≥ 10 mg/L.
* Unequivocal cranial symptoms of GCA (new-onset localized headache, scalp or temporal artery tenderness, ischemia-related vision loss, or otherwise unexplained mouth or jaw pain upon mastication) AND/OR symptoms of polymyalgia rheumatica (PMR) defined as shoulder and/or hip girdle pain associated with inflammatory morning stiffness
* Temporal artery biopsy revealing features of GCA AND/OR
* evidence of large-vessel vasculitis by angiography or cross-sectional imaging study such as magnetic resonance angiography (MRA), computed tomography angiography (CTA), positron emission tomography-computed tomography (PET CT), or ultrasound

Patients with new onset GCA or relapsing GCA (Definition new onset: diagnosis of GCA within 6 weeks of Baseline Visit; Definition relapsing GCA: diagnosis of GCA (in accordance with inclusion criterion no. 4) > 6 weeks before Baseline Visit and in the meantime achieved remission (absence of signs and symptoms attributable to GCA and normalization of ESR (< 30 mm/hr) and CRP (<10.0mg/L) included) including previous treatment with ≥ 25 mg/day prednisolone equivalent for ≥ 2 weeks.)

Active disease as defined by the presence of signs and symptoms of GCA (cranial or PMR) and elevated ESR ≥ 30 mm/hr, or CRP ≥ 10 mg/L, attributed to active GCA within 6 weeks of Baseline.

Prednisolone dose of 25-60 mg/day at Baseline.

Exclusion Criteria:

Previous exposure to secukinumab or other biologic drug directly targeting Interleukin(IL)-17 or IL-17 receptor.

Patients treated with any cell-depleting therapies including but not limited to anti-CD20 or investigational agents (e.g. anti-CD3, anti-CD4, anti-CD5 or anti-CD19).

Patients who have previously been treated with any biologic agent including but not limited to tocilizumab, sirukumab, abatacept, or tumor necrosis factor alpha (TNFα) inhibitors (infliximab, adalimumab, etanercept, certolizumab, golimumab).

Patients who have previously been treated with tofacitinib or baricitinib.

Patients treated with i.v. immunoglobulins or plasmapheresis within 8 weeks prior to Baseline.

Patients treated with cyclophosphamide, tacrolimus or everolimus within 6 months prior to Baseline.

Patients treated with hydroxychloroquine, cyclosporine A, azathioprine, sulfasalazine or mycophenolate mofetil within 4 weeks of Baseline.

Patients treated with leflunomide within 8 weeks of Baseline unless a cholestyramine washout has been performed in which case the patient must be treated within 4 weeks of Baseline.

Patients treated with an alkylating agent except for cyclophosphamide as mentioned above.

Patients requiring systemic chronic glucocorticoid therapy for any other reason than GCA.

Chronic systemic glucocorticoid therapy over the last 4 years or longer; or inability, in the opinion of the investigator, to withdraw glucocorticoid therapy through protocol-defined taper regimen due to suspected or established adrenal insufficiency.

Patients requiring chronic (i.e. not occasional "prn") high potency opioid analgesics for pain management.

Active ongoing inflammatory diseases or underlying metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions, which in the opinion of the investigator immunosuppressed the patient and/or places the patient at unacceptable risk for participation in an immunomodulatory therapy.

History of renal trauma, glomerulonephritis, or patients with one kidney only, or a serum creatinine level exceeding 1.8 mg/dL (159.12 μmol/L).

Screening total white blood cell (WBC) count < 3000/μL, or platelets < 100 000/μL or neutrophils < 1500/μL or hemoglobin < 8.3 g/dL (83 g/L).

Major ischemic event, unrelated to GCA, within 12 weeks of screening.

Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C at screening or randomization.

Life vaccinations within 6 weeks prior to Baseline or planned vaccination during study participation until 12 weeks after last study treatment administration.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Germany (11):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Germering
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Venhoff N, Schmidt WA, Bergner R, Rech J, Unger L, Tony HP, Finzel S, Andreica I, Kofler DM, Weiner SM, Lamprecht P, Schulze-Koops H, App C, Pournara E, Mendelson MH, Sieder C, Maricos M, Thiel J. Safety and efficacy of secukinumab in patients with giant cell arteritis (TitAIN): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Rheumatol. 2023 Jun;5(6):e341-e350. doi: 10.1016/S2665-9913(23)00101-7. PMID 38251601
- [Derived] Venhoff N, Schmidt WA, Lamprecht P, Tony HP, App C, Sieder C, Legeler C, Jentzsch C, Thiel J. Efficacy and safety of secukinumab in patients with giant cell arteritis: study protocol for a randomized, parallel group, double-blind, placebo-controlled phase II trial. Trials. 2021 Aug 17;22(1):543. doi: 10.1186/s13063-021-05520-1. PMID 34404463
- See also: Clinical_Trials_Results_Word_Form-CAIN457ADE11C.docx attachment has been refreshed from the Clinical Trials Results Word Form template. Data may be populated from the following (as available) : Study (70.0), Protocol (4.22), Results(0.22) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217151&parentIdentifier=CAIN457ADE11C&attachmentIdentifier=99008743-0238-47ae-a207-9328edbb241c&fileName=Clinical_Trials_Results_Word_Form-CAIN457ADE11C.docx&versionIdentifier=
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 11 investigative sites in 1 country.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations were performed up to 6 weeks before the beginning of the Treatment period.
Period: Overall Study
Arm/Group | Secukinumab | Placebo
Started | 27 | 25
Completed | 22 | 17
Not Completed | 5 | 8
Not completed — Subject decision | 2 | 3
Not completed — Physician Decision | 2 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned by randomization and who received at least one dose of randomized study treatment (secukinumab or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.4 (5.31) | 69.6 (8.02) | 73.1 (7.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 10 | 7 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Sustained Remission Until Week 28
Description: Remission was defined as the absence of flare. Sustained remission was defined as the absence of flare until Week 28 and in adherence to the protocol prednisolone taper regimen.
  Flare was determined by the investigator and was defined as the recurrence after remission of signs or symptoms of Giant Cell Arteritis (GCA) and/or erythrocyte sedimentation rate (ESR) greater than or equal to (>/=) 30 millimeters per hour (mm/hr) and/or C-reactive Protein (CRP) (>/=10.0 mg/L) attributable to GCA.
  Patients were classified as non-responders if they did not achieve remission within 12 weeks of Baseline (remission referred to the absence of flare), were in the "escape arm" (this referred to patients entering escape between Baseline and Week 28), prematurely discontinued study treatment prior to Week 28 (absence of flare was checked prior to study treatment administration), did not have information to evaluate sustained remission response until Week 28.
Time Frame: Until week 28
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 25
Participants | 19 | 6
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Odds Ratio; Test type: Superiority; Odds Ratio (OR) = 9.31, 95% CI 2-sided [3.54 to 26.29] — Odd Ratio (posterior median) median and 95% credibility interval calculated using the Bayesian inference

2. Secondary Outcome: Percentage of Participants in Remission at Week 12
Description: Remission was defined as the absence of flare. Sustained remission was defined as the absence of flare until Week 28 and in adherence to the protocol prednisolone taper Regimen.
  Flare was determined by the investigator and was defined as the recurrence after remission of signs or symptoms of GCA and/or erythrocyte sedimentation rate (ESR) greater than or equal to (>/=) 30 millimeters per hour (mm/hr) and/or CRP (>/=10.0 mg/L) attributable to GCA.
  Patients were classified as non-responders if they did not achieve remission within 12 weeks of Baseline (remission referred to the absence of flare), were in the "escape arm" (this referred to patients entering escape between Baseline and Week 28), prematurely discontinued study treatment prior to Week 28 (absence of flare was checked prior to study treatment administration), did not have information to evaluate sustained remission response until Week 28.
Time Frame: Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 25
Participants | 22 | 12

3. Secondary Outcome: Time to First GCA Flare After Clinical Remission
Description: Flare was determined by the investigator and was defined as the recurrence after remission of signs or symptoms of GCA and/or erythrocyte sedimentation rate (ESR) greater than or equal to (>/=) 30 millimeters per hour (mm/hr) and/or CRP (>/=10.0 mg/L) attributable to GCA. Time to first flare after remission referred to time from first day of study treatment until first post-Baseline flare.
  For time to first GCA flare after remission (up to and including Week 52), patients who prematurely discontinued study treatment prior to Week 52 were censored at the time of premature discontinuation and patients who completed treatment and did not have a flare were censored at their last visit in the treatment phase.
  Time to first GCA flare after remission was calculated using Kaplan-Meier plot of time.
Time Frame: Up to Week 52 (included)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 25
days | NA [NA to NA] — NA: not enough participants with events to calculate the median & CI | 197.0 [101.0 to 280.0]

4. Secondary Outcome: Total Cumulative Prednisolone Dose Over 28 Weeks and 52 Weeks
Description: Total cumulative co-administered prednisolone treatment was summarized over time by treatment arm. Patients received a daily dose of prednisolone, which was decreased (i.e. tapered down) from Baseline to Week 26. No additional prednisolone or equivalent was permitted.
Time Frame: from Baseline to week 28, from baseline to week 52 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 25
milligrams
  Baseline to Week 28 | 2689.70 (935.860) | 2693.74 (1241.907)
  Baseline to Week 52 | 2841.26 (1116.192) | 3375.58 (1720.978)

5. Secondary Outcome: Percentage of Participants With GCA Who Had Sustained Remission Until Week 52
Description: Remission was defined as the absence of flare. Sustained remission was defined as patients without flare until Week 52 and in adherence to the protocol prednisolone taper regimen plus prednisolone-free phase from Week 27 onwards. Flare was determined by the investigator and was defined as the recurrence after remission of signs or symptoms of GCA and/or erythrocyte sedimentation rate (ESR) greater than or equal to (>/=) 30 millimeters per hour (mm/hr) and/or CRP (>/=10.0 mg/L) attributable to GCA.
  Patients were classified as non-responders if they did not achieve remission within 12 weeks of Baseline (remission referred to the absence of flare), were in the "escape arm" (this referred to patients entering escape between Baseline and Week 28), prematurely discontinued study treatment prior to Week 28 (absence of flare was checked prior to study treatment administration), did not have information to evaluate sustained remission response until Week 28.
Time Frame: Until Week 52
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 25
Participants | 16 | 2

6. Secondary Outcome: Number of Participants on Prednisolone Dose ≤ 5mg/Day
Description: Number of participants on co-administered prednisolone treatment ≤ 5mg/day who responded at Week 19, Week 26 and Week 52.
  Remission was defined as the absence of flare. Sustained remission was defined as the absence of flare until Week 28 and in adherence to the protocol prednisolone taper Regimen. There were 2 taper regimens: for patients on 40 to 60 mg/day prednisolone at Baseline and for patients on 25 to 40 mg/day prednisolone at Baseline depending on patients' prednisolone levels at Baseline. Prednisolone was tapered from a dose of 25 mg to 60 mg at Baseline to 1 mg at Week 26 [last dose].
Time Frame: Week 19, Week 28, Week 52
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned by randomization and who received at least one dose of randomized study treatment (secukinumab or placebo). n represents the number of participants with a value for a specific categorical variable at Week 19, 28 and 52.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 25
Participants
  Week 19 (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 19 (n = 25, 20) | 22 | 10
  Week 28 (n = 23, 20): number analyzed (Participants) | 23 | 20
  Week 28 (n = 23, 20) | 19 | 9
  Week 52 (n = 21, 17): number analyzed (Participants) | 21 | 17
  Week 52 (n = 21, 17) | 19 | 13

7. Secondary Outcome: Physicians Global Assessment (PhGA) of Disease Activity: Change From Baseline Score Via Visual Analogue Scale (VAS)
Description: Clinician Reported Outcome: Physicians global assessment (PhGA) using a visual analogue scale (VAS) scale. VAS is a range of scores from 0-100, with lower change from baseline scores indicating a more favorable outcome and higher change from baseline scores indicating a greater disease activity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 36, 44 & 52
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment had been assigned by randomization and who received at least one dose of randomized study treatment (secukinumab or placebo). The change from baseline at each visit is calculated only for subjects with a value at baseline and the particular visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 23
scores on a scale
  Week 4 (n = 27, 23) | -4.8 (14.43) | -3.2 (18.45)
  Week 8 (n = 26, 21): number analyzed (Participants) | 26 | 21
  Week 8 (n = 26, 21) | -5.8 (12.77) | 2.1 (18.94)
  Week 12 (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12 (n = 25, 20) | -3.4 (21.93) | -3.1 (10.81)
  Week 16 (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16 (n = 25, 20) | -4.1 (15.62) | 0.7 (13.97)
  Week 20 (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20 (n = 24, 20) | -6.9 (14.78) | -1.5 (14.32)
  Week 24 (n = 23, 20): number analyzed (Participants) | 23 | 20
  Week 24 (n = 23, 20) | -4.3 (15.92) | 2.2 (17.22)
  Week 28 (23, 19): number analyzed (Participants) | 23 | 19
  Week 28 (23, 19) | -5.4 (15.61) | 3.9 (21.47)
  Week 36 (21, 19): number analyzed (Participants) | 21 | 19
  Week 36 (21, 19) | -8.7 (18.45) | 0.7 (17.45)
  Week 44 (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44 (n = 21, 16) | -5.5 (16.87) | 1.1 (15.20)
  Week 52 (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52 (n = 21, 16) | -9.5 (16.72) | 4.0 (21.24)

8. Secondary Outcome: Patients Global Assessment (PGA) of Disease Activity: Change From Baseline Via Visual Analogue Scale (VAS)
Description: Patient Reported Outcome: Patients global assessment (PGA) score using a VAS scale. VAS is a range of scores from 0-100, with lower change from baseline scores indicating a more favorable outcome and higher change from baseline scores indicating a greater disease activity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 36, 44 & 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 23
scores on a scale
  Week 4 (n = 27, 23) | -15.8 (28.17) | -0.5 (23.58)
  Week 8 (n = 26, 21): number analyzed (Participants) | 26 | 21
  Week 8 (n = 26, 21) | -15.8 (27.61) | -10.8 (27.64)
  Week 12 (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12 (n = 25, 20) | -8.0 (29.43) | -11.9 (31.46)
  Week 16 (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16 (n = 25, 20) | -18.6 (19.39) | -8.8 (31.43)
  Week 20 (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20 (n = 24, 20) | -19.18 (30.68) | -6.9 (31.94)
  Week 24 (n = 23, 20): number analyzed (Participants) | 23 | 20
  Week 24 (n = 23, 20) | -14.9 (28.84) | -7.0 (30.61)
  Week 28 (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28 (n = 23, 19) | -14.4 (25.46) | -8.0 (31.31)
  Week 36 (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36 (n = 21, 19) | -20.9 (22.31) | -8.6 (29.90)
  Week 44 (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44 (n = 21, 16) | -21.7 (27.35) | -9.4 (30.58)
  Week 52 (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52 (n = 21, 16) | -19.2 (27.35) | -15.9 (24.04)

9. Secondary Outcome: Change From Baseline in FACIT-Fatigue Scale
Description: Patient Reported Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue is a 13-item questionnaire with a full scale of 0 -52 that assesses self-reported fatigue and its impact upon daily activities and function. The higher the score the better functioning (less fatigue).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 36, 44 & 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 23
scores on a scale
  Week 4 (n = 27, 23) | 2.11 (9.613) | -0.96 (7.358)
  Week 8 (n = 26, 21): number analyzed (Participants) | 26 | 21
  Week 8 (n = 26, 21) | 2.19 (10.190) | 0.81 (7.498)
  Week 12 (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12 (n = 25, 20) | 0.96 (11.175) | -0.25 (10.047)
  Week 16 (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16 (n = 25, 20) | 2.12 (8.876) | -0.36 (8.884)
  Week 20 (n =24, 20): number analyzed (Participants) | 24 | 20
  Week 20 (n =24, 20) | 3.42 (8.617) | 0.05 (10.318)
  Week 24 (n = 23, 20): number analyzed (Participants) | 23 | 20
  Week 24 (n = 23, 20) | 2.91 (10.409) | -3.10 (11.281)
  Week 28 (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28 (n = 23, 19) | 3.61 (11.044) | 0.42 (9.203)
  Week 36 (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36 (n = 21, 19) | 3.90 (7.245) | 1.84 (8.719)
  Week 44 (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44 (n = 21, 16) | 2.67 (5.986) | 0.31 (10.928)
  Week 52 (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52 (n = 21, 16) | 3.19 (7.033) | 0.19 (8.848)

10. Secondary Outcome: Change From Baseline in Short-Form (SF)-36 Questionnaire
Description: Patient Reported Outcome: The SF-36 is a standardized questionnaire used to measure health-related quality of life among healthy patients and patients with acute and chronic conditions. It consists of 8 subscales that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. The higher the score (change from baseline) the more favorable the outcome. The values were reported by change from baseline in SF-36 domain scores.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 36, 44 & 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 23
scores on a scale
  Week 4: Physical Functioning (PF) (n = 27, 23) | 0.14 (7.562) | -1.25 (4.417)
  Week 8: PF (n = 26 ,21): number analyzed (Participants) | 26 | 21
  Week 8: PF (n = 26 ,21) | -0.44 (8.849) | 0.18 (4.987)
  Week 12: PF (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12: PF (n = 25, 20) | 0.38 (6.322) | -0.38 (8.750)
  Week 16: PF (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16: PF (n = 25, 20) | -0.00 (8.646) | -0.86 (6.814)
  Week 20: PF (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20: PF (n = 24, 20) | 0.80 (8.098) | -0.10 (6.495)
  Week 24: PF (n = 22, 20): number analyzed (Participants) | 22 | 20
  Week 24: PF (n = 22, 20) | 0.52 (5.702) | -2.11 (8.667)
  Week 28: PF (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28: PF (n = 23, 19) | 1.25 (5.276) | -0.40 (6.460)
  Week 36: PF (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36: PF (n = 21, 19) | 1.37 (5.778) | -1.31 (6.631)
  Week 44: PF (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44: PF (n = 21, 16) | 1.00 (6.674) | -0.36 (8.065)
  Week 52: PF (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52: PF (n = 21, 16) | 2.46 (4.770) | 0.12 (5.696)
  Week 4: Role-Physical (R-P) (n =27, 23) | 3.49 (7.886) | 0.49 (10.616)
  Week 8: R-P (n =26, 21): number analyzed (Participants) | 26 | 21
  Week 8: R-P (n =26, 21) | 3.80 (9.628) | -0.75 (10.515)
  Week 12: R-P (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12: R-P (n = 25, 20) | 3.32 (9.3301) | 1.01 (9.539)
  Week 16: R-P (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16: R-P (n = 25, 20) | 4.58 (8.947) | -1.12 (8.847)
  Week 20: R-P (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20: R-P (n = 24, 20) | 4.40 (9.538) | -0.45 (8.163)
  Week 24: R-P (n = 22, 20): number analyzed (Participants) | 22 | 20
  Week 24: R-P (n = 22, 20) | 3.37 (7.458) | -0.00 (10.094)
  Week 28: R-P (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28: R-P (n = 23, 19) | 5.96 (10.034) | 1.77 (8.553)
  Week 36: R-P (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36: R-P (n = 21, 19) | 5.99 (6.444) | 0.24 (10.121)
  Week 44: R-P (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44: R-P (n = 21, 16) | 5.13 (6.515) | 0.70 (11.262)
  Week 52: R-P (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52: R-P (n = 21, 16) | 6.20 (6.659) | 1.40 (9.126)
  Week 4: Bodily Pain (BP) (n = 27, 23) | 8.03 (13.272) | 7.68 (11.235)
  Week 8: BP (n = 26, 21: number analyzed (Participants) | 26 | 21
  Week 8: BP (n = 26, 21 | 5.80 (14.475) | 9.68 (10.485)
  Week 12: BP (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12: BP (n = 25, 20) | 6.92 (13.426) | 6.84 (11.674)
  Week 16: BP (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16: BP (n = 25, 20) | 7.69 (14.841) | 4.50 (13.560)
  Week 20: BP (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20: BP (n = 24, 20) | 6.10 (14.072) | 8.63 (12.457)
  Week 24: BP (n = 22, 20): number analyzed (Participants) | 22 | 20
  Week 24: BP (n = 22, 20) | 5.97 (12.689) | 3.93 (11.952)
  Week 28: BP (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28: BP (n = 23, 19) | 6.47 (12.643) | 6.32 (13.149)
  Week 36: BP (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36: BP (n = 21, 19) | 7.20 (13.724) | 7.81 (10.794)
  Week 44: BP (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44: BP (n = 21, 16) | 8.01 (15.378) | 9.00 (7.910)
  Week 52: BP (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52: BP (n = 21, 16) | 5.49 (12.328) | 8.39 (11.866)
  Week 4: General Health (GH) ( n = 27, 23) | 3.49 (9.207) | 0.23 (6.761)
  Week 8: GH (n = 26, 21): number analyzed (Participants) | 26 | 21
  Week 8: GH (n = 26, 21) | 2.74 (8.119) | 0.18 (6.758)
  Week 12: GH (n = 25, 20: number analyzed (Participants) | 25 | 20
  Week 12: GH (n = 25, 20 | 2.22 (7.383) | 0.62 (8.158)
  Week 16: GH (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16: GH (n = 25, 20) | 2.28 (8.235) | -0.74 (7.858)
  Week 20: GH (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20: GH (n = 24, 20) | 4.50 (6.774) | -0.38 (7.933)
  Week 24: GH (n = 22, 20): number analyzed (Participants) | 22 | 20
  Week 24: GH (n = 22, 20) | 2.85 (7.149) | -0.19 (9.031)
  Week 28: GH (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28: GH (n = 23, 19) | 3.53 (7.285) | 1.18 (7.837)
  Week 36:GH (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36:GH (n = 21, 19) | 3.42 (6.680) | -0.47 (7.833)
  Week 44: GH (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44: GH (n = 21, 16) | 1.02 (8.127) | -0.30 (9.597)
  Week 52: GH (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52: GH (n = 21, 16) | 3.03 (6.733) | 0.15 (10.277)
  Week 4: Vitality (n = 27, 23) | 4.07 (8.607) | -1.42 (7.699)
  Week 8: Vitality (n = 26, 21): number analyzed (Participants) | 26 | 21
  Week 8: Vitality (n = 26, 21) | 2.17 (7.952) | 0.71 (8.185)
  Week 12: Vitality (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12: Vitality (n = 25, 20) | 3.57 (7.477) | -0.30 (9.241)
  Week 16: Vitality (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16: Vitality (n = 25, 20) | 4.28 (7.431) | -0.45 (7.847)
  Week 20: Vitality (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20: Vitality (n = 24, 20) | 4.70 (8.445) | 0.45 (9.652)
  Week 24: Vitality (n = 22, 20): number analyzed (Participants) | 22 | 20
  Week 24: Vitality (n = 22, 20) | 3.78 (7.112) | -1.93 (11.697)
  Week 28: Vitality (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28: Vitality (n = 23, 19) | 6.20 (7.489) | 0.16 (6.679)
  Week 36: Vitality (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36: Vitality (n = 21, 19) | 7.07 (7.060) | 1.41 (5.635)
  Week 44: Vitality (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44: Vitality (n = 21, 16) | 6.08 (8.375) | -0.93 (12.497)
  Week 52: Vitality (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52: Vitality (n = 21, 16) | 7.21 (8.690) | 0.37 (11.474)
  Week 4: Social Functioning (SF) (n = 27, 23) | 3.71 (7.939) | 1.74 (7.499)
  Week 8: SF (n = 26, 21): number analyzed (Participants) | 26 | 21
  Week 8: SF (n = 26, 21) | 4.82 (8.327) | 2.63 (9.979)
  Week 12: SF (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12: SF (n = 25, 20) | 4.01 (9.154) | 1.76 (7.325)
  Week 16: SF (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16: SF (n = 25, 20) | 5.21 (11.069) | 0.75 (7.325)
  Week 20: SF (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20: SF (n = 24, 20) | 4.81 (10.080) | 3.51 (8.150)
  Week 24: SF (n = 22, 20): number analyzed (Participants) | 22 | 20
  Week 24: SF (n = 22, 20) | 4.56 (8.602) | 0.00 (10.912)
  Week 28: SF (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28: SF (n = 23, 19) | 3.49 (8.476) | 3.17 (9.631)
  Week 36: SF (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36: SF (n = 21, 19) | 7.16 (10.703) | 5.01 (7.285)
  Week 44: SF (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44: SF (n = 21, 16) | 6.45 (8.988) | 0.63 (11.561)
  Week 52: SF (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52: SF (n = 21, 16) | 7.16 (8.621) | 2.82 (9.681)
  Week 4: Role-Emotional (RE) (n = 27, 23) | -0.77 (12.454) | 3.48 (12.985)
  Week 8: RE (n = 26, 21): number analyzed (Participants) | 26 | 21
  Week 8: RE (n = 26, 21) | 3.08 (11.457) | 1.99 (13.239)
  Week 12: RE (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12: RE (n = 25, 20) | -0.42 (12.076) | 0.52 (13.188)
  Week 16: RE (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16: RE (n = 25, 20) | 3.76 (10.586) | -0.00 (11.465)
  Week 20: RE (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20: RE (n = 24, 20) | 3.48 (11.058) | 0.35 (11.569)
  Week 24: RE (n = 22, 20): number analyzed (Participants) | 22 | 20
  Week 24: RE (n = 22, 20) | 2.85 (11.753) | -1.22 (16.025)
  Week 28: RE (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28: RE (n = 23, 19) | 3.63 (11.853) | 1.10 (11.725)
  Week 36: RE (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36: RE (n = 21, 19) | 5.47 (10.066) | 0.73 (16.518)
  Week 44: RE (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44: RE (n = 21, 16) | 4.15 (12.293) | 3.26 (16.354)
  Week 52: RE (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52: RE (n = 21, 16) | 6.14 (11.385) | 0.43 (19.234)
  Week 4: Mental Health (MH) (n = 27, 23) | 3.0 (8.514) | 0.57 (8.420)
  Week 8: MH (n = 26, 21): number analyzed (Participants) | 26 | 21
  Week 8: MH (n = 26, 21) | 2.82 (10.643) | 1.49 (6.950)
  Week 12: MH (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 12: MH (n = 25, 20) | 3.14 (10.786) | 4.45 (7.690)
  Week 16: MH (n = 25, 20): number analyzed (Participants) | 25 | 20
  Week 16: MH (n = 25, 20) | 4.29 (8.337) | 5.36 (6.379)
  Week 20: MH (n = 24, 20): number analyzed (Participants) | 24 | 20
  Week 20: MH (n = 24, 20) | 3.49 (10.926) | 6.41 (7.984)
  Week 24: MH (n = 22, 20): number analyzed (Participants) | 22 | 20
  Week 24: MH (n = 22, 20) | 2.62 (8.730) | 2.61 (13.149)
  Week 28: MH (n = 23, 19): number analyzed (Participants) | 23 | 19
  Week 28: MH (n = 23, 19) | 2.84 (9.816) | 6.06 (7.350)
  Week 36: MH (n = 21, 19): number analyzed (Participants) | 21 | 19
  Week 36: MH (n = 21, 19) | 5.98 (8.111) | 5.64 (8.988)
  Week 44: MH (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 44: MH (n = 21, 16) | 4.11 (8.969) | 1.14 (11.891)
  Week 52: MH (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52: MH (n = 21, 16) | 5.73 (7.473) | 4.25 (11.257)

11. Secondary Outcome: Change From Baseline in EQ-5D-5L (EuroQol 5D) Questionnaire
Description: EQ-5D-5L, a self-administered questionnaire assessing health status in adults, is divided into 2 sections. The 1st section addresses 5 dimensions (mobility, self-care, usual activity, pain/discomfort, & anxiety/depression). Items are rated either "no problem", "slight problems", "moderate problems", "severe problems", or "extreme problems/unable." A composite health index is defined by combining the levels for each dimension. The 2nd section measures self-rated (global) health status via vertically oriented VAS where 100 represents the "best possible health state" & 0 represents the "worst possible health state." The EQ-5D-5L contains 6 items assessing health status via a single index value or health utility score and allows "weighting" by the patient of health states & generation of patient utilities. Published weights are available allowing for creation of a single summary health utility score. Scores range from 0 to 1, with lower scores representing a higher level of dysfunction.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 36, 44 & 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 27 | 23
scores on a scale
  EQ-5D-5L VAS: Week 4 (n = 27, 23) | 11.26 (16.819) | 1.87 (21.467)
  EQ-5D-5L VAS: Week 8 (n = 26, 21): number analyzed (Participants) | 26 | 21
  EQ-5D-5L VAS: Week 8 (n = 26, 21) | 5.58 (16.650) | 5.52 (29.646)
  EQ-5D-5L VAS: Week 12 (n = 25, 20): number analyzed (Participants) | 25 | 20
  EQ-5D-5L VAS: Week 12 (n = 25, 20) | 4.64 (19.598) | 3.30 (22.850)
  EQ-5D-5L VAS: Week 16 (n = 25, 20): number analyzed (Participants) | 25 | 20
  EQ-5D-5L VAS: Week 16 (n = 25, 20) | 7.000 (19.530) | 4.40 (27.354)
  EQ-5D-5L VAS: Week 20 (n = 24, 20): number analyzed (Participants) | 24 | 20
  EQ-5D-5L VAS: Week 20 (n = 24, 20) | 7.88 (19.077) | 6.30 (25.041)
  EQ-5D-5L VAS: Week 24 (n = 23, 20): number analyzed (Participants) | 23 | 20
  EQ-5D-5L VAS: Week 24 (n = 23, 20) | 5.39 (17.598) | -1.00 (29.902)
  EQ-5D-5L VAS: Week 28 (n = 23, 19): number analyzed (Participants) | 23 | 19
  EQ-5D-5L VAS: Week 28 (n = 23, 19) | 4.43 (17.840) | 10.37 (21.670)
  WEQ-5D-5L VAS: Week 36 (n = 21, 19): number analyzed (Participants) | 21 | 19
  WEQ-5D-5L VAS: Week 36 (n = 21, 19) | 6.90 (17.972) | 5.32 (28.825)
  EQ-5D-5L VAS: Week 44 (n = 21, 16): number analyzed (Participants) | 21 | 16
  EQ-5D-5L VAS: Week 44 (n = 21, 16) | 6.38 (19.505) | 12.69 (21.941)
  EQ-5D-5L VAS: Week 52 (n = 21, 16): number analyzed (Participants) | 21 | 16
  EQ-5D-5L VAS: Week 52 (n = 21, 16) | 11.62 (16.877) | 10.81 (24.109)
  EQ-5D-5L utility index: Week 4 (n = 27, 23) | 0.0166 (0.19559) | -0.0702 (0.21239)
  EQ-5D-5L utility index: Week 8 (n = 26, 21): number analyzed (Participants) | 26 | 21
  EQ-5D-5L utility index: Week 8 (n = 26, 21) | -0.0034 (0.19972) | 0.0087 (0.9869)
  EQ-5D-5L utility index: Week 12 (n = 25, 20): number analyzed (Participants) | 25 | 20
  EQ-5D-5L utility index: Week 12 (n = 25, 20) | 0.0016 (0.16236) | -0.0122 (0.15686)
  EQ-5D-5L utility index: Week 16 (n = 25, 20): number analyzed (Participants) | 25 | 20
  EQ-5D-5L utility index: Week 16 (n = 25, 20) | 0.0186 (0.14639) | -0.0196 (0.19789)
  EQ-5D-5L utility index: Week 20 (n = 24, 20): number analyzed (Participants) | 24 | 20
  EQ-5D-5L utility index: Week 20 (n = 24, 20) | 0.0210 (0.13308) | 0.0221 (0.16759)
  EQ-5D-5L utility index: Week 24 (n = 23, 20): number analyzed (Participants) | 23 | 20
  EQ-5D-5L utility index: Week 24 (n = 23, 20) | 0.0402 (0.12427) | -0.0444 (0.20875)
  EQ-5D-5L utility index: Week 28 (n = 23, 19): number analyzed (Participants) | 23 | 19
  EQ-5D-5L utility index: Week 28 (n = 23, 19) | -0.0002 (0.06695) | 0.0240 (0.13458)
  EQ-5D-5L utility index: Week 36 (n = 21, 19): number analyzed (Participants) | 21 | 19
  EQ-5D-5L utility index: Week 36 (n = 21, 19) | 0.0063 (0.06432) | -0.0155 (0.13186)
  EQ-5D-5L utility index: Week 44 (n = 21, 16): number analyzed (Participants) | 21 | 16
  EQ-5D-5L utility index: Week 44 (n = 21, 16) | -0.0119 (0.08525) | 0.0090 (0.13033)
  EQ-5D-5L utility index: Week 52 (n = 21, 16): number analyzed (Participants) | 21 | 16
  EQ-5D-5L utility index: Week 52 (n = 21, 16) | -0.0076 (0.11997) | 0.0205 (0.09403)

12. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. This was assessed in order to identify the presence of inflammation, to determine its severity, and to monitor response to treatment. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
Time Frame: Baseline, Week 28, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 23 | 18
mm/hr
  Week 28 (n = 23, 18) | 4.043 (16.1934) | 14.667 (23.9141)
  Week 52 (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52 (n = 21, 16) | -3.286 (10.6167) | 10.000 (14.8728)

13. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) Level
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. This was assessed in order to identify the presence of inflammation, to determine its severity, and to monitor response to treatment. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 28, Week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 23 | 19
mg/L
  Week 28 (n = 23, 19) | 4.426 (9.6836) | 5.216 (8.9820)
  Week 52 (n = 21, 16): number analyzed (Participants) | 21 | 16
  Week 52 (n = 21, 16) | -1.433 (8.7909) | 4.650 (14.3691)

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from first dose of study treatment and co-administered Prednisolone treatment until end of treatment (48 weeks) plus 4 weeks (52 weeks). The mean/standard deviation exposure to the study treatment was 49.5 (9.6) weeks for secukinumab and 46.9 (12.6) weeks for placebo. The mean/standard deviation exposure to the co-administered prednisolone treatment was 307 (9.6) weeks for secukinumab and 43.2 (12.2) weeks for placebo.
Description: Adverse Event (AE): Any sign or symptom that occurs during treatment plus 30 days post treatment.
Groups:
- All Participants: All participants who participated in the study.
Arm/Group | Secukinumab | Placebo | All Participants
All-Cause Mortality (participants affected / at risk) | 1/27 | 1/25 | 2/52
Serious Adverse Events (participants affected / at risk) | 6/27 | 11/25 | 17/52
Other Adverse Events (participants affected / at risk) | 25/27 | 23/25 | 48/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=27) | Placebo (N=25) | All Participants (N=52)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 2
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 1
Noninfective sialoadenitis (Gastrointestinal disorders) | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Inflammatory marker increased (Investigations) | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 1
Neurological symptom (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=27) | Placebo (N=25) | All Participants (N=52)
Cushingoid (Endocrine disorders) | 1 | 2 | 3
Glaucoma (Eye disorders) | 2 | 2 | 4
Vision blurred (Eye disorders) | 1 | 2 | 3
Dental caries (Gastrointestinal disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 4
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Fatigue (General disorders) | 2 | 1 | 3
Oedema peripheral (General disorders) | 2 | 4 | 6
Gastroenteritis (Infections and infestations) | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 5 | 5 | 10
Oral candidiasis (Infections and infestations) | 4 | 1 | 5
Respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Rhinitis (Infections and infestations) | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 4 | 2 | 6
Bone contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2 | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Blood pressure increased (Investigations) | 0 | 2 | 2
C-reactive protein increased (Investigations) | 1 | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Dizziness (Nervous system disorders) | 3 | 0 | 3
Headache (Nervous system disorders) | 4 | 3 | 7
Polyneuropathy (Nervous system disorders) | 2 | 0 | 2
Sciatica (Nervous system disorders) | 1 | 2 | 3
Tension headache (Nervous system disorders) | 1 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Giant cell arteritis (Vascular disorders) | 1 | 2 | 3
Haematoma (Vascular disorders) | 1 | 3 | 4
Hypertension (Vascular disorders) | 6 | 8 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e. data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT03765788/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT03765788/SAP_001.pdf